CLINICAL TRIAL: NCT00037791
Title: Safety and Efficacy of (PN-152,243)/PN-196,444 in the Prevention of Thrombocytopenia in Patients Receiving Myelosuppressive Treatment Regimens Requiring Platelet Transfusion Support.
Brief Title: Safety and Efficacy of (PN-152,243)/PN-196,444 in the Prevention of Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 98-OTPO-005
Record Dates: First submitted 2002-05-21; First posted 2002-05-22 (Estimated); Last update posted 2006-11-09 (Estimated); Status verified 2006-09

CONDITIONS: Neoplasms; Thrombocytopenia; Multiple Myeloma; Lymphoma, Malignant
MeSH Terms: conditions — Neoplasms; Thrombocytopenia; Multiple Myeloma; Lymphoma

INTERVENTIONS:
Drug: (PN-152,243)/PN-196,444

SUMMARY:
Intensive chemotherapy is associated with significant thrombocytopenia, often requiring platelet transfusion to maintain platelet counts. This investigational drug has demonstrated the ability to increase platelet counts. This study will test the safety and efficacy of this investigational drug in the prevention of thrombocytopenia in patients with solid tumors, lymphomas or multiple myeloma who are receiving myelosuppressive treatment regimens requiring platelet transfusion support.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have solid tumors, lymphomas or multiple myeloma who are receiving myelosuppressive treatment regimens requiring platelet transfusion support

Exclusion Criteria:

* Patients must not have active bleeding (exclusions do apply) or history of platelet disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 1999-12; Study Completion 2002-09

PRIMARY OUTCOMES:
To evaluate the effectiveness of two schedules of intravenous rhTPO versus placebo as secondary prophylaxis in reducing the proportion of patients requiring platelet transfusion for severe chemotherapy-induced thrombocytopenia.

SECONDARY OUTCOMES:
Identify the effect of rhTPO on the number of episodes of severe chemotherapy-induced thrombocytopenia(platelet count <15,000/mm3) and the number of platelet transfusions
Evaluate the severity and duration of thrombocytopenia and neutropenia associated with rhTPO Prophylaxis
Quantify the effect of rhTPO on the occurrence of any bleeding events associated with thrombocytopenia
Assess the likelihood that patients will have adequate hematologic recovery to allow on-time chemotherapy administration in the subsequent cycle
Assess the safety of multiple intravenous doses of rhTPO
Determine the occurrence and clinical implications of any anti-rhTPO antibodies
Evaluate the impact of rhTPO prophylaxis on health economics/cost effectiveness
Evaluate the impact of rhTPO administration on patient quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (5):
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Houston, Texas
- Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D., Argentina
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=98-OTPO-005&StudyName=Safety+and+Efficacy+of+%28PN%2D152%2C243%29%2FPN%2D196%2C444+in+the+Prevention+of+Thrombocytopenia+